CLINICAL TRIAL: NCT05299593
Title: 24-hour Efficacy and Tolerability of the Tafluprost-timolol Fixed Association Without Preservatives in Glaucomatous or Ocular Hypertensive Patients Already Treated With Latanoprost Preserved With BAK. A Prospective, Open Study of 3 Months Duration.
Acronym: HERO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HERO
Record Dates: First submitted 2022-02-15; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-02

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: Glaucoma, ocular hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — tafluprost; Timolol

STUDY DESIGN:
Intervention Model Description: Single group, open label
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tafluprost/timolol (Experimental): Enrolled patients will be treated with one drop of the fixed combination Tafluprost-Thymol without preservative in the evening at 20.00 (+/- 1 hour). Patients will be administrered with one drop in the conjunctival sac of the affected eye (s) once a day.
  Interventions: Drug: tafluprost/timolol

INTERVENTIONS:
Drug: tafluprost/timolol — One ml active drug contains: 15 micrograms of tafluprost and 5 mg of timolol (as maleate).
  A single-dose container (0.3 ml) of eye drops, solution, contains 4.5 micrograms of tafluprost and 1.5 mg of timolol. One drop (about 30 µl) contains about 0.45 micrograms of tafluprost and 0.15 mg of timolol. Patients will be administrered with one drop in the conjunctival sac of the affected eye (s) once a day.

SUMMARY:
This is a phase IV, interventional, multi-center, open clinical Trial. Patients will be administered one eye drop of tafluprost/timolol fixed combination at 20:00 (+/- 1 hour), in the treatment of open angle glaucoma and ocular hypertension. The patients will suspend the treatment with latanoprost.

DETAILED DESCRIPTION:
This is a phase IV, interventional, multi-center, not comparative, open clinical Trial to evaluate the effectiveness in reducing the mean 24-hour IOP of the preservative-free fixed combination of Tafluprost 0.0015% and Timolol 0.5% administered once at night (8pm) in POAG or OHT patients suffering from mild OSD and requiring further IOP reduction while in topical treatment with BAK-preserved Latanoprost 0.05 mg/ml. Three Italian recruiting centers are included in the study and the estimated number of patients to be enrolled is 43. After evaluating the patient's eligibility, the patients will suspend the treatment with latanoprost and will be administered one eye drop of tafluprost/timolol fixed combination at 20:00 (+/- 1 hour) at the end of the V1B visit. Active drug will be contained (about 30 µl, one drop) contains about 0.45 micrograms of tafluprost and 0.15 mg of timolol.

The Study consists in 6 Visits:

1. Screening visit V0 and baseline V1A.
2. Treatment period visit V1B; V2; V3A; V3B.
3. End of study V3B.

ELIGIBILITY:
Inclusion Criteria:

1. Ocular hypertension or primary open-angle glaucoma or secondary to dispersion of pigment or pseudoesfoliatio;
2. IOP <22 mmHg in latanoprost therapy in both eyes since at least 6 weeks and > 17 mmHg in at least one eye;
3. OSD at least mild as defined by DEQ-5 (score> 6);
4. Examination of the visual field during the three months prior to enrollment (if not present, the patient must be subjected to a visual field at the screening visit);
5. Treatment with latanoprost BAK-preserved from at least 6 weeks;
6. Subject agrees to follow the study procedures and signs the EC-approved ICF;
7. For women of child-bearing potential, blood screening for beta-HCG before randomization and use of one effective method of birth control during the conduct of the study

Exclusion Criteria:

1. Inability to understand and sign informed consent;
2. Age under 18 years;
3. Other forms of secondary glaucoma (besides pigmentary and pseudoesfoliatius);
4. Narrow angle or history of acute glaucoma attacks;
5. Previous history of trabeculoplasty in the previous 6 months;
6. History of glaucoma surgery or refractive surgery;
7. Cataract surgery in the 6 months prior to enrollment;
8. Contraindications to the use of beta-blockers (reactive airway disease, including bronchial asthma or a history of bronchial asthma, severe chronic obstructive pulmonary disease; sinus bradycardia, sick sinus syndrome, including sinoatrial block, second or third degree atrioventricular block not controlled by pacemaker; full-blown heart failure, cardiogenic shock);
9. Damage to the visual field with a mean deviation (MD) <-20 dB;
10. BCVA <2/10;
11. Topical ocular drugs performed within 3 months prior to enrollment that may interfere with the study results (eg steroids, non-steroidal anti-inflammatory drugs, immunosuppressants, etc.);
12. Use of tear substitutes containing preservatives within 30 days prior to enrollment;
13. Any other condition that, in the opinion of the investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful completion of the study or would impair interpretation of results;
14. Corneal anomalies that preclude an accurate measurement of IOP (eg astigmatism> 3 D, keratoconus, opacity or corneal ulcers);
15. Any type of previous corneal or conjunctival surgery including pterygium removal or refractive surgery;
16. Unstable systemic disorders that may require the initiation or variation of therapies that may influence intraocular pressure during the study;
17. Woman of childbearing potential, or who is currently pregnant or breastfeeding;
18. Inability to adhere to the procedures required by the protocol or to the studio treatment;
19. Participation in another experimental therapeutic protocol within one month prior to baseline and during the study period (participation in natural history study is allowed);
20. Hypersensitivity to the active substances or to any of the excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
The evaluation of the mean 24-h absolute Intraocular Pressure (IOP) | through study completion, an average of 3 months
  Reduction measured in mmHg (millimeters of mercury).

SECONDARY OUTCOMES:
Evaluation of the average reduction of Intraocular Pressure(IOP) at 24-hour | through study completion, an average of 3 months
  Curve measured in mmHg.
Evaluation of the percentage reduction of the average Intraocular Pressure(IOP) of the 24 hours | through study completion, an average of 3 months
  percentage at each time point.
Evaluation of the average daytime reduction and night of the Intraocular Pressure(IOP) | through study completion, an average of 3 months
  Measured in mmHg
Evaluation of the percentage of patients achieving Intraocular Pressure(IOP) reduction in average | through study completion, an average of 3 months
  reductions in average IOP at 24h when plus 20%, when plus 25%,when plus 30%.
Evaluation of the changes in the Corneale Staining Test (CFS) and Break-up Time Test (tBUT) parameters | through study completion, an average of 3 months
  with fluorescein, measured area and density
Evaluation of the changes in Dry Eye Questionnaire (DEQ-5) | through study completion, an average of 3 months
  DEQ-5 questionnaire Score
Evaluation of the changes of the number, activation of corneal, conjunctival dendritic cells to confocal microscopy. | through study completion, an average of 3 months
  Changes number corneal and dendritic cells
Evaluation of the changes of the number of conjunctival goblet cells to confocal microscopy | through study completion, an average of 3 months
  Changes of number of goblet cells
Evaluation of the changes in quality of life | through study completion, an average of 3 months
  NEIVFQ-25 questionnaire (score).

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Oddone, MD, Principal Investigator — IRCCS G.B.Bietti Foundation for the study and Research in Ophthalmology ONLUS; Luciano Quaranta, MD, Principal Investigator — Università di Pavia Policlinico S. Matteo; Luca Rossetti, MD, Principal Investigator — ASST Santi Paolo e Carlo
Locations (3):
- Italy (3):
  - ASST Santi Paolo e Carlo, Milan
  - Università di Pavia Policlinico S. Matteo, Pavia
  - IRCCS G.B.Bietti Foundation for the study and Research in Ophthalmology ONLUS, Roma

IPD SHARING:
Plan to Share IPD: No
There is not a Plan to make available to other researches.